CLINICAL TRIAL: NCT03451812
Title: Molecular PET/MR Imaging in Vivo Validation of Biomarker for Human Prostate Cancer
Acronym: PCAPETMR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Gigin Lin, Associate Professor, Chang Gung Memorial Hospital
Other Study IDs: 105-6435C; 104-4855A (Other: CGMH)
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Prostate Adenocarcinoma
Keywords: prostate cancer; metabolomics; molecular imaging; PET; MRI; 11C-choline tracer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Device: No

GROUPS / COHORTS (1):
- prostate cancer: The newly diagnostic number for the high-risk PCa patients in our hospital annually is ~70, it is clinically feasible to recruit 40 patients a year since the study begins. The study could be completed in 3 years with 120 cases.

SUMMARY:
Primary objective:

To correlate the blood/urine metabolomic biomarkers with PET/MR imaging.

Secondary objectives:

1. To evaluate the sensitivity and specificity of the PET/MR in diagnosis of prostate cancer.
2. To examine the diagnostic performance among subgroups of defined high-risk and low-risk subjects.
3. To interrogate the metabolomic alterations with the molecular PET/MR to develop workable panel biomarkers.

DETAILED DESCRIPTION:
According to 2015 National Comprehensive Cancer Network (NCCN) guideline, medical imaging plays important roles for detection and staging for PCa, in addition to blood or urine biomarkers. Although there are a number of very different diagnostic imaging methods, e.g. transrectal ultrasound (TRUS), computed tomography (CT), magnetic resonance (MR) imaging and spectroscopy, or 18F-FDG positron emission tomography (PET), none of these have gained a dominant role as the optimum method for all clinical scenarios.The recently added armamentarium, PET/MR, might improve diagnosis in this regard.

Therefore, we conduct this trial to identify the ability of [11C]Choline PET/MR to evaluate the patients with prostate cancer, especially under the circumstance of elevated PSA level.

ELIGIBILITY:
Inclusion Criteria:

* Males
* 40-85 years of age
* Patients with a biopsy-proven or clinically highly suspected prostate adenocarcinoma, or benign prostatic hyperplasia
* Able to tolerate [11C]Choline PET scan and MRI scan
* Written informed consent from the patient

Exclusion Criteria:

* Acute prostatitis or non-urologic bacterial infection requiring medical treatment within the last 3 months.
* History of AIDS in the period prior to the screening.3
* Contraindications to [11C]Choline PET/MR scans

  1. Surgical implants including pacemaker implants, cochlear implants, dentures held in place by magnets imbedded in the gums and aneurysm clips except those inserted at CGMH
  2. Metallic prosthesis of the hip or pelvic region
  3. Renal function impairment with estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73 m2
  4. Claustrophobia
  5. Medical drugs with choline
  6. Previous allergy to carbon-labeled radionuclide
* Active other malignancy within the last 2 years
* Subject which in the opinion of the investigator preclude participation for scientific reasons, for reasons of compliance, or for reasons of the subject's safety.
* Prisoners or patients with mental illness

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in a tertiary referral center.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy | 1 year
  sensitivity, specificity, accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Gigin Lin, MD, PhD, Principal Investigator — Medical Imaging and Intervention, Chang Gung Memorial Hospital
Locations (1):
- Department of Medical Imaging and Intervention, Chang Gung Memorial Hospital, Guishan, Taoyuan, Taiwan